CLINICAL TRIAL: NCT01071304
Title: A Study to Evaluate the Effect of Multiple Doses of Ridaforolimus (AP23573; MK-8669) on the Single Dose Pharmacokinetics of Midazolam.
Brief Title: Effect of Ridaforolimus on the Pharmacokinetics of Midazolam (Study MK-8669-044)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-044; 2010_511
Record Dates: First submitted 2010-02-17; First posted 2010-02-19 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Relapsed or Refractory Advanced Cancer
Keywords: Relapsed or refractory advanced cancer, metastatic cancer, locally advanced cancer
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis | interventions — Midazolam; ridaforolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): In Part 1, all participants received a single oral dose of 2 mg midazolam on Day -2. On Days 1-5, all participants received daily single oral doses of ridaforolimus 40 mg ( 4 x 10 mg tablets). On Day 5, all participants received a single oral dose of 2 mg midazolam coadministered with the dose of ridaforolimus. Participants had the option to continue into Part 2 of this study.
  Interventions: Drug: Midazolam; Drug: Ridaforolimus

INTERVENTIONS:
Drug: Midazolam — A single oral dose of midazolam 2 mg (1 mL of 2 mg/mL syrup) was given on Day -2 and Day 5.
Drug: Ridaforolimus — Ridaforolimus 40 mg (4 x 10 mg tablets) oral once daily on Days 1 through 5.

SUMMARY:
The purpose of this study is to compare the pharmacokinetic profile of midazolam given alone and midazolam given after multiple oral doses of 40 mg ridaforolimus.

Part 1 of this study is designed for evaluating CYP3A4 activity following 5 days of dosing of ridaforolimus and is not designed with efficacy endpoints. Part 2 is a compassionate-use extension to give patients an opportunity to receive a clinically active dose of ridaforolimus. Part 2 dosing is open ended with limited data collection.

ELIGIBILITY:
Inclusion Criteria:

* participant is male or female
* participant must have a histologically or cytologically-confirmed metastatic or locally

advanced solid tumor, lymphoma, or hematologic malignancy that has failed to

respond to standard therapy, progressed despite standard therapy, or for which

standard therapy does not exist. There is no limit on the number of prior treatment

regimens

* participant must have a performance status of ≤ 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* If participant is female she must be post menopausal (defined as free from menses for ≥1

year and follicle stimulating hormone (FSH) is in the postmenopausal range at screening), surgically sterilized

(hysterectomy, oophorectomy or tubal ligation) or, if of childbearing potential, must

be willing to use 2 approved methods of contraception (hormonal contraception,

intra-uterine device, diaphragm with spermicide, cervical cap with spermicide or

female condom with spermicide; spermicides alone are not an acceptable method of

contraception) from screening until 30 days following the last dose of study drug.

* If participant is female and of childbearing potential, she must have a negative serum β-

human chorionic gonadotropin (hCG) pregnancy test at screening and within 24 hrs prior to dosing Part 1/Day -2

* If participant is male and has female partner(s) of child-bearing potential, he must agree

to use a medically acceptable method of contraception during the study and for 30

days after the last dose of study drug. If the participant's partner is pregnant, the participant

must agree to use a condom. If the participant's partner is of child-bearing potential, he

must use a condom and his partner must additionally use one of the following

methods: hormonal contraception, intra-uterine device, diaphragm with spermicide,

cervical cap with spermicide or female condom with spermicide.

- participant must have laboratory values within the parameters as outlined in the study protocol.

* participant has a life expectancy of >3 months.
* participant has voluntarily agreed to participate by giving written informed consent.

Inclusion Criteria for Part 2 of the study:

* participant has enrolled in and complied with study procedures in Part 1 of the study.
* participant is willing to comply with protocol requirements and procedures for Part 2 of

the study.

Exclusion Criteria:

- participant has had chemotherapy, radiotherapy, or biological therapy within 4 weeks (6

weeks for nitrosoureas, mitomycin C, and monoclonal antibodies) prior to first dose

of study drug (Part 1/Day -2) or who has not recovered from adverse events due to

agents administered more than 4 weeks earlier.

* participant is receiving any other concurrent anti-cancer therapy; participant may be receiving supportive therapy as defined in the study protocol
* participant is receiving concurrent treatment with immunosuppressive agents, including

corticosteroids at doses greater than those used for replacement therapy. Corticosteroids administered for replacement therapy at stable doses for ≥ 2 weeks are permitted.

- participant has clinically significant abnormality on electrocardiogram (ECG) performed

at the prestudy (screening) visit and/or prior to administration of the initial dose of

study drug.

- participant has significant or uncontrolled cardiovascular disease or a history of

congestive heart failure, unstable angina, or myocardial infarction. Controlled

hypertension < 150/100 mm Hg is allowed if participant is on a stable antihypertensive

regimen.

- participant is currently participating or has participated in a study with an investigational

compound or device within 30 days prior to the first dose of study drug.

- participant has a primary central nervous system tumor, an active brain metastases or

leptomeningeal carcinomatosis. participants with previously treated brain metastases that

are stable for > 3 months are eligible if a current brain magnetic resonance imaging (MRI) (within 28 days of the first dose of study drug) shows no edema or evidence of progression compared to a

prior MRI study (≥ 3 months ago).

- participant has a history or current evidence of any condition, therapy, or lab abnormality

that might confound the results of the study, interfere with the participant's participation

for the full duration of the study, or is not in the best interest of the participant to

participate.

- participant has a known psychiatric disorder that would interfere with giving informed

consent or cooperating with the requirements of the study.

- participant is, at the time of signing informed consent, a regular user (including

use of any illicit drugs or had a recent history (within the last year) of

drug or alcohol abuse.

- participant is pregnant or breastfeeding, or expecting to conceive within the projected

duration of the study.

* participant is known to be Human Immunodeficiency Virus (HIV)-positive.
* participant has a known history of Hepatitis B or C.
* participant has newly diagnosed (within 3 months before the first dose of study drug) or

poorly controlled Type 1 or 2 diabetes.

- participant requires treatment with medications that are inducers or inhibitors of

cytochrome P450 (CYP3A) prior to the first dose of study drug (Part 1/Day -2) and throughout the study until the

poststudy visit.

- participant is currently taking or has a history of pronounced sedation upon taking

benzodiazepine or other sedative/soporific. The washout from prestudy use of these

medications should be at least five half-lives prior to the first dose of study drug in

Part 1 (Part 1/Day -2) and use during Part 1 is not permitted (use in Part 2 is

permitted).

- participant has an active infection or has received intravenous antibiotics, antiviral, or

antifungal agents within 2 weeks prior to the first dose of the study drug.

- participant will not refrain from the use of herbal remedies (such as St. John's Wort,

shark cartilage, etc.) from 2 weeks prior to the first dose (Part 1/Day -2) and

throughout the duration of the study.

- participant is anticipated to require immunologic therapy, radiation therapy, surgery, or

chemotherapy during the study.

* participant has received high-dose chemotherapy with stem cell rescue.
* participant has had a blood transfusion within one week of study entry.
* participant is unable to swallow capsules and/or has a documented surgical or anatomical

condition that will preclude the participant from swallowing and absorbing oral

medications on an ongoing basis.

- participant has a known hypersensitivity to the components of the study drug or its

analogs or macrolide antibiotics (e.g., clarithromycin, erythromycin, azithromycin).

* participant has an allergy or hypersensitivity to midazolam or other benzodiazepines.
* participant will not refrain from consumption of grapefruit or grapefruit juice for

approximately 2 weeks prior to first dosing (Part 1/Day -2) until the completion of the

study.

- participant has not adequately recovered from any prior surgical procedure or has

undergone any major surgical procedure within 4 weeks prior to the first dose of

study drug. participants who have undergone minor procedures (e.g. placement of a

central venous access port) will be considered eligible it they have fully recovered.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve (AUC [0-infinity]) of midazolam 2 mg administered alone versus when administered after multiple oral doses of ridaforolimus 40 mg. | 8 days (Day -2 through Day 5, 24 hrs postdose)
Maximum Concentration (Cmax) of midazolam 2 mg administered alone versus when administered after multiple oral doses of ridaforolimus 40 mg. | 8 days (Day -2 through Day 5, 24 hrs postdose)
Time to Cmax (Tmax) of a single oral dose of 2 mg midazolam administered alone versus when administered after multiple oral doses of ridaforolimus 40 mg. | 8 days (Day -2 through Day 5, 24 hrs postdose)
Apparent terminal half-life (t½) of a single oral dose of 2 mg midazolam administered alone versus when administered after multiple oral doses of ridaforolimus 40 mg. | 8 days (Day -2 through Day 5, 24 hrs postdose)

REFERENCES:
- [Result] Stroh M, Talaty J, Sandhu P, McCrea J, Patnaik A, Tolcher A, Palcza J, Orford K, Breidinger S, Narasimhan N, Panebianco D, Lush R, Papadopoulos KP, Wagner JA, Trucksis M, Agrawal N. Lack of meaningful effect of ridaforolimus on the pharmacokinetics of midazolam in cancer patients: model prediction and clinical confirmation. J Clin Pharmacol. 2014 Nov;54(11):1256-62. doi: 10.1002/jcph.331. Epub 2014 May 24. PMID 24827931